CLINICAL TRIAL: NCT03161262
Title: SMS-Based Follow-Ups to Improve Post-Discharge Surgical Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Rondi Gelbard, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00094000
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Surgical Site Infection
Keywords: Text-message reminder; Post-operative medication; Behavioral Research; Social Research; Short Message Service (SMS)
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either the intervention group or control group. The test group constitutes receiving consistent medication reminders, as per the patient's prescribed frequency, and weekly surveys prompting them to report their pain level and an image of their surgical site for the duration of the full 3 months. The control group will not receive medication reminders or questions regarding their pain or surgical site. Both control and test groups will receive a monthly questionnaire via SMS to assess patient satisfaction with the intervention and changes in medication adherence behaviors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS-based reminders (Experimental): This group will receive consistent medication reminders, as per the patient's prescribed frequency, and weekly surveys prompting them to report their pain level and an image of their surgical site. They will also receive a monthly questionnaire via SMS to assess patient satisfaction with the intervention and changes in medication adherence behaviors.
  Interventions: Behavioral: SMS-based reminders
- Control group (No Intervention): The control group will not receive medication reminders or questions regarding their pain or surgical site. This group will receive a monthly questionnaire via SMS to assess patient satisfaction with the intervention and changes in medication adherence behaviors.

INTERVENTIONS:
Behavioral: SMS-based reminders — The SMS-based reminders consist of sending messages to participants assigned to this study arm reminding them to take their medication and prompting participants to complete surveys. Medication reminders are sent as per the participant's prescribed frequency and weekly surveys allow participants to report their pain level as well as send an image of their surgical site. Beyond pre-determined reminders and surveys sent to patients, the Memora Health platform is interactive and allows patients to text in questions they may have regarding their medications, care, or condition. Participants will receive the messages for 3 months.
  Other Names: Memora Health platform
  Arms: SMS-based reminders

SUMMARY:
The purpose of this study is to determine whether low-cost Short Message Service (SMS)-based follow-up medication reminders and surveys for surgical site infection (SSI) reporting can improve outcomes by increasing medication adherence and earlier detection and care of SSI. This will be a prospective study involving enrollment of patients onto the Memora Health platform, a web application developed for automating SMS content to patients. Post-operative patients will be identified by providers and enrolled prior to discharge, after which they will be followed for 3 months.

Primary endpoints include medication adherence and patient satisfaction with the text messaging tool. Secondary endpoints include early detection of SSIs, patient satisfaction with overall post-discharge care and health-related quality of life, and pertinent 30-day readmissions.

DETAILED DESCRIPTION:
Post-operative follow up with patients is critical to providing high quality and cost effective care. In the current standard of care, patients receive verbal instructions from their physician along with discharge paperwork that outlines best practices for self-care. Unfortunately, difficult instructions can be miscommunicated or be overwhelming, and patients often leave confused, resulting in poor patient care post-discharge and high 30-day readmission rates. Medication adherence represents a crucial area for follow-up, as it is a major determinant of high-quality outcomes for post-operative care. Specifically, over 50% of patients in the U.S. either forget to or don't correctly take their prescription medications. Non-adherence causes nearly 10% of all hospital admissions in the U.S. and 125,000 annual deaths.

In a survey of 10,000 patients, the most common reported reason for missing medications was forgetfulness (24%), followed by perceived side effects (20%), high drug costs (17%), and perception that a prescribed medication would have little effect on their disease (14%). The majority of the factors contributing to non-adherence could therefore be resolved by longitudinally addressing forgetfulness and misconceptions about medication effectiveness, options for treatment, and side effects.

An SMS patient engagement case-management platform (Memora Health, Boston, MA) has been created that enables providers to input a new medication regimen into a web-based, HIPAA compliant app that then sends text message reminders to the patient to take their medication. Communication is two-way, therefore not only helping to improve adherence and self-management for the patient, but also providing care staff with more data on the post-discharge behavior and care satisfaction of their patients. While the value of SMS-based interventions on health outcomes is abundant in the literature, there is a paucity of data evaluating the impact of SMS follow-up on improving surgical outcomes through improved medication adherence and early detection of SSI. The purpose of this study is to utilize Memora Health, a platform that leverages mobile messaging as a medium for advancing preventive care, to improve the quality of post-operative care delivered to patients, and thereby improve patient satisfaction as well as reducing readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a working cell phone that can send and receive SMS/Multimedia Messaging Service (MMS) over the next three months
* Patient has a working cell phone with a camera
* Being able to read and write fluently in English
* All patients identified in the Electronic Medical Record (EMR) with International Classification of Diseases (ICD)-10 codes for patients who underwent procedures with external wounds and can be at risk of surgical site infection (SSI). Only patients falling under the categories of 'Major Diagnostic' and 'Major Therapeutic' will be considered.

Exclusion Criteria:

* Patient deceased prior to discharge
* Patient transferred to another hospital
* Patient has a terminal illness with less than 3-month expected survival
* Vulnerable populations including patients who are in the middle of a pregnancy or prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Medication adherence assessed with patient responses to medication reminders | Month 3
  Overall patient response rates to SMS reminders will be used to assess medication compliance. Participants are asked to reply to the reminders when they have taken the dose of medication.
Medication adherence assessed by Adherence to Refills and Medications Survey (ARMS) | Month 3
  The Adherence to Refills and Medications Survey (ARMS-7) is a 7-item survey asking respondents about their medication-taking behavior and factors that contribute to medication compliance or non-compliance. Participants select a score for each question ranging from 1-4, where 1 represents 'None' and 4 represents 'All'. The scores are treated as a continuous measure, with total points being added up, with lower scores indicating high adherence and high scores indicating low adherence.
Participant Satisfaction | Month 1 through Month 3
  Patient satisfaction with the SMS tool will be assessed using a 7-item survey administered at the conclusion of the study. Participants will rate the message reminders on a scale from 1 (very poor) to 5 (very good): helpfulness, ease of use, ease of understanding, frequency of messages, quality of messages, likelihood of continuing to use message reminders, and willingness to recommend message reminders to a friend.

SECONDARY OUTCOMES:
Early detection of surgical site infection (SSI) | Month 3
  Participants will be allowed to intermittently provide pain scores and pictures of their surgical sites to help increase early detection of surgical site infection (SSI) post-discharge. The value of these images in early detection of SSIs will be measured through physician reporting of SSIs.
Early intervention of surgical site infection (SSI) | Month 3
  Participants will be allowed to intermittently provide pain scores and pictures of their surgical sites to help increase early detection of surgical site infection (SSI) post-discharge. The number of incidents of early intervention for SSIs will be determined as a method of measuring early detection of SSIs.
Care Transitions Measure (CTM-15) Score | Day 1, Month 3
  Care Transitions Measure (CTM-15) is a 15-item survey asking respondents to indicate their degree of agreement with statements relating to the quality of care transition from being hospitalized to being discharged. Respondents select from: 1=Strongly Disagree, 2=Disagree, 3=Agree, 4=Strongly Agree. Missing responses and selections of "Don't Know/Don't Remember/Not Applicable" do not contribute to the total score. A mean score is obtained and higher scores indicate a better transition during hospital discharge.
Number of visits with provider | Day 1, Month 3
  Responses to the question "In the last 3 months, how many times did you visit this provider to get care for yourself?" will be compared between study groups.
Number of appointments for routine care | Day 1, Month 3
  Responses to the question "In the last 3 months, did you make any appointments for a check-up or routine care with this provider? (1 = yes, 2 = no)" will be compared between study groups.
Satisfaction with time spent by provider on care | Day 1, Month 3
  Responses to the question "In the last 3 months, did the provider spend enough time on your care?" will be compared between study groups. Participants rate their satisfaction with the amount of time their provider spent on their care on a 5-point scale where 1 = strongly agree and 5 = strongly disagree.
Overall rating of provider | Day 1, Month 3
  Responses to the question "Using any number from 0 to 10, where 0 is the worst provider possible and 10 is the best provider possible, what number would you use to rate this provider?" will be compared between study groups.
30-Day Readmission | Day 30
  Readmission to the hospital within 30 days of hospital discharge will be obtained through Electronic Health Records. Any hospital admissions will be analyzed to determine if they are related to the recent procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Rondi B Gelbard, MD, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided